CLINICAL TRIAL: NCT05713305
Title: Effect of an Online Self-help Psychological Intervention on the Physical and Mental Health of Non-professional Staff Who Supported the ICU During the Omicron Outbreak: a Randomized Controlled Trial
Brief Title: Effect of an Online Self-help Psychological Intervention on Non-ICU Specialty Care During the COVID-19 Outbreak
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-0023
Record Dates: First submitted 2023-01-18; First posted 2023-02-06 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2023-01

CONDITIONS: SARS-CoV-2 Infection; Staff Attitude; Anxiety; Mental Health Issue
MeSH Terms: conditions — COVID-19; Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Daily members of the intervention group were thought to provide three different forms of daily sessions each day, averaging 10-20 minutes. These sessions included psycho-educational and cognitive-behavioral exercises, music therapy, sleep hygiene, stress relief methods. Weekly online lecture sessions presented by professional mental health therapists. In-depth interviews are conducted both before and after the experiment to explore the feasibility of the intervention
  Interventions: Procedure: Online-based self-help psychological intervention
- Control group (Placebo Comparator): They will receive official mental health recommendations on how to cope mentally with the pandemic. These recommendations inform about the importance of a daily structure, social contact, acceptance of negative emotions and strengthening of positive emotions, and stimulus control to assimilate SARS-CoV-2 Omicron-related news. In-depth interviews are conducted both before and after the experiment to explore the feasibility of the intervention
  Interventions: Procedure: Provide online mental health knowledge

INTERVENTIONS:
Procedure: Online-based self-help psychological intervention — Daily members of the intervention group were thought to provide three different forms of daily sessions each day, averaging 10-20 minutes. These sessions included psycho-educational and cognitive-behavioral exercises, music therapy, sleep hygiene, stress relief methods. Weekly online lecture sessions presented by professional mental health therapists
  Arms: Intervention group
Procedure: Provide online mental health knowledge — They will receive official mental health recommendations on how to cope mentally with the pandemic. These recommendations inform about the importance of a daily structure, social contact, acceptance of negative emotions and strengthening of positive emotions, and stimulus control to assimilate SARS-CoV-2 Omicron-related news
  Arms: Control group

SUMMARY:
Timely interventions may reduce the occurrence of post-traumatic stress disorder (PTSD) in ICU medical staff. Existing research suggests that either self-learning psychological relief methods or seeking online counseling or therapy from professional psychotherapists during the SARS-CoV-2 Omicron outbreak has the potential to alleviate the emotional distress and promote the physical and mental health of health care workers. Web-based online mental health interventions complemented by joint effective mental health advice can further reduce harmful negative effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Non-ICU professional staff providing direct health care services to critically ill SARS-CoV-2 Omicron patients in the ICU
3. Signing the informed consent form

Exclusion Criteria:

1. No reported acute suicidal tendencies
2. No history of psychotic or dissociative symptoms
3. Pregnancy or lactation
4. Major family changes within the last 12 weeks( For e.g. death of immediate family member)
5. Participated in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Changes in medical staff DASS-21( Depression Anxiety Stress Scale 21) after 28 days of intervention | 28 days after intervention
  DASS-21 changes( 0-63), The larger the score, the worse the result

SECONDARY OUTCOMES:
Proportion of depression and anxiety problems among different types of staff | 28 days after intervention
  Proportion of depression and anxiety
The degrees to which depression and anxiety problems occur in different types of staff | 28 days after intervention
  The degrees to which depression and anxiety problems
Incidence of posttraumatic stress disorder | 28 days after intervention
  Incidence of posttraumatic stress disorder
Well-being was measured with the WHO-5 well-being index | 28 days after intervention
  Well-being was measured with the WHO-5 well-being index ( 0-25), The higher the score, the higher the happiness index
Improvement in sleep quality | 28 days after intervention
  Improvement in sleep quality( ISI), insomnia severity index ( 0-28) , The larger the score, the worse the result
Results of the Depression Anxiety Stress Scale 21 scale after 3 months of intervention | Three months after intervention
  DASS-21 changes( 0-63), The larger the score, the worse the result ，after three months of intervention
Results of the Depression Anxiety Stress Scale 21 scale after 6 months of intervention | 6 months after intervention
  DASS-21 changes( 0-63), The larger the score, the worse the result， after 6 months of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided